CLINICAL TRIAL: NCT01035554
Title: Effect of a Novel Behavioral Intervention on Blood Pressure Control in Hypertension Patients
Brief Title: Behavioral Study to Control Blood Pressure
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Milton S. Hershey Medical Center (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Christopher Sciamanna, MD, MPH, Principal Investigator, Milton S. Hershey Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 687; R01HL089402-01A2 (NIH)
Record Dates: First submitted 2009-12-17; First posted 2009-12-18 (Estimated); Last update posted 2013-11-11 (Estimated); Status verified 2013-11

CONDITIONS: Hypertension
Keywords: high blood pressure
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Usual Care (UC) + Printed Materials (PM) (Active Comparator): If the participant is assigned to UC, they will receive standard care. They will not receive a HBPM to use for the study, but will be given one to keep at the 3 month Follow-Up Visit. If they are also assigned to PM, they will then be given written materials (pamphlets from the NIH) and will be asked to review the information in its entirety. The coordinator will be available to answer any questions they might have.
  Interventions: Other: Usual Care; Other: Printed Materials
- UC + Self-Paced Program Instruction (SPPI) (Experimental): If the participant is assigned to UC, they will receive standard care. They will not receive a HBPM to use for the study, but will be given one to keep at the 3 month Follow-Up Visit. If they are also assigned to SPPI, they will be asked to complete a series of educational modules at their own pace on the laptop that is provided. They will be informed that there is no grading and that the program is set up so that they can go at their own pace. The SPPI modules will be designed directly from the information provided on the Printed Materials from the National Institutes of Health.
  Interventions: Other: Self-Paced Programmed Instruction (SPPI); Other: Usual Care
- Home Blood Pressure Monitor (HBPM) + PM (Experimental): If the participant is assigned to HBPM, they will be asked to use the monitor once a day in the morning and once before they go to bed any 3 days of the week, each week of the study (total = 12 weeks). They will be asked to record their BP values in diaries they will be given to take home with them. If they are also assigned to PM, they will then be given written materials (pamphlets from the NIH) regarding hypertension education and will be asked to review the information in its entirety. The coordinator will be available to answer any questions they might have.
  Interventions: Other: Home Blood Pressure Monitor; Other: Printed Materials
- HBPM + SPPI (Experimental): If the participant is assigned to HBPM, they will be asked to use the monitor once a day in the morning and once before they go to bed any 3 days of the week, each week of the study (total = 12 weeks). They will be asked to record their BP values in diaries they will be given to take home with them.
  If they are also assigned to SPPI, they will be asked to complete a series of educational modules at their own pace on the laptop that is provided. They will be informed that there is no grading and that the program is set up so that they can go at their own pace. The SPPI modules will be designed directly from the information provided on the PM from the National Institutes of Health.
  Interventions: Other: Self-Paced Programmed Instruction (SPPI); Other: Home Blood Pressure Monitor

INTERVENTIONS:
Other: Self-Paced Programmed Instruction (SPPI) — If participants are assigned to SPPI, they will be asked to complete a series of educational modules at their own pace on the laptop that is provided. They will be informed that there is no grading and that the program is set up so that they can go at their own pace. The SPPI modules will be designed directly from the information provided on the Printed Materials (PM) from the National Institutes of Health.
  Arms: HBPM + SPPI; UC + Self-Paced Program Instruction (SPPI)
Other: Home Blood Pressure Monitor — The home blood pressure monitor will allow the participant to measure their blood pressure anytime and anywhere precisely, quickly and easily on their upper arm.
  Other Names: Carrera Upper Arm Blood Pressure Monitor (battery opperated)
  Arms: HBPM + SPPI; Home Blood Pressure Monitor (HBPM) + PM
Other: Usual Care — Standard care
  Arms: UC + Self-Paced Program Instruction (SPPI); Usual Care (UC) + Printed Materials (PM)
Other: Printed Materials — National Institutes of Health Printed Materials on hypertension
  Other Names: NIH publications 96-4041, 4042, 4045, 4046, 4047
  Arms: Home Blood Pressure Monitor (HBPM) + PM; Usual Care (UC) + Printed Materials (PM)

SUMMARY:
We propose to test an intervention to increase patients' understanding of the causes, consequences, and the rationale for treatment, of their hypertension (HTN), as a strategy for increasing blood pressure (BP) control. The focus is on the interaction between a behavioral intervention to reduce BP - home BP monitoring (HBPM) - and patient knowledge, which, we propose, moderates the effect of the HBPM intervention. We hypothesize that patients who have a better understanding of their illness and its prescribed treatment will be more adherent to the treatment regimen, and thus will exhibit improved outcomes compared to those who have been exposed to the same intervention, but who do not have a clear understanding of these elements.

DETAILED DESCRIPTION:
According to the National Health and Nutrition Examination Survey, more than 31% of adults in the U.S. population have hypertension (HTN). HTN is a major risk factor for heart disease and stroke, which are the 1st and 3rd leading causes of death in the U.S. and impose an enormous financial and social burden on Americans with more than $352 billion spent in direct and indirect costs. Behavioral interventions to control blood pressure (BP) have exhibited, on average, positive but relatively modest effects on blood pressure control. We and others have studied the effects of one such intervention - home BP monitoring - on BP control in hypertensive patients, and found reliable, albeit modest effects. We have found similar effects for another behavioral intervention, Motivational Interviewing, on BP control. We hypothesize that the effects of such interventions will be augmented when accompanied by a systematic approach to patient education concerning their illness and its treatment. The literature suggests that patient education is "necessary but not sufficient"(an implicit interaction) to produce behavioral changes; however, the "necessary" part tends to be ignored by interventionalists. The implication of the interaction is that when patients lack the necessary knowledge, any intervention is likely to be less effective (as any value multiplied by zero - i.e., no knowledge - is zero). In spite of this, we have found no trials that have tested the interaction between patient knowledge and a lifestyle or drug intervention.

We propose to test an intervention to increase patients' understanding of the causes, consequences, and the rationale for treatment, of their HTN, as a strategy for increasing BP control. The focus is on the interaction between a behavioral intervention to reduce BP - home BP monitoring (HBPM) - and patient knowledge, which, we propose, moderates the effect of the HBPM intervention. We hypothesize that patients who have a better understanding of their illness and its prescribed treatment will be more adherent to the treatment regimen, and thus will exhibit improved outcomes compared to those who have been exposed to the same intervention, but who do not have a clear understanding of these elements.

We propose to pilot test the effect of the HBPM intervention using a 2 X 2 independent groups randomized design, to allow us to compare the effects of Usual Care (UC) + Printed Materials (PM) compared to Usual Care (UC) and Self-Paced Programmed Instruction (SPPI) compared to Home Blood Pressure Monitoring (HBPM) + Printed Materials (PM) compared to Home Blood Pressure Monitoring (HBPM) + Self-Paced Programmed Instruction (SPPI).

Our primary hypothesis is:

Decreased ABP at 3 months will be ordered thusly:

HBPM+SPPI > HBPM+PM > UC+SPPI > UC+PM

ELIGIBILITY:
Inclusion Criteria:

* English speaking
* Has been diagnosed by physician has having hypertension/high blood pressure
* Has been prescribed medications to treat hypertension
* Has a blood pressure reading at the Screening Visit of either above 140/90
* If previously diagnosed with cancer, must be in remission
* Not currently pregnant or trying to become pregnant within next three months
* No major kidney, heart, liver failure
* Ages 21-80
* Must be able to travel to Hershey Medical Center (Hershey, PA)

Exclusion Criteria:

* Cannot read and speak English fluently
* Has not been diagnosed with hypertension
* Is not currently taking medications for hypertension
* Has blood pressure that is below 140 and 90
* Has blood pressure that is above 180 or 120
* Has cancer that is not in remission
* Is currently pregnant of plans to become pregnant in the next 3 months
* Has had major kidney, heart or liver failure
* Is less than 21 or greater than 80 years old

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 203 (Actual)
Dates: Start 2010-05; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Decreased Arterial Blood Pressure | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Sciamanna, MD, MPH, Principal Investigator — Milton S. Hershey Medical Center
Locations (1):
- Penn State Hershey Medical Center, Hershey, Pennsylvania, United States